CLINICAL TRIAL: NCT05626075
Title: Correlation Between Corneal Topographic Patterns and Refractive Status Of The Eye in Sohag City,Egypt
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Abdallah Abdelaal, Ophthalmology Resident at Akhemim Central hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Soh-Med-22-07-2014
Record Dates: First submitted 2022-10-12; First posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Eye Change
Keywords: Topographic; visual acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group Low Myopia (Experimental): 1. Patients with low myopia aging more than 15 years old
  2. All patients are with visual acuity (uncorrected, with habitual correction, and best spectacle correction).
  3. There is no restrictions on the range and regularity of keratometry
  Interventions: Diagnostic Test: Using Oculus Pentacam® which is s a rotating Scheimpflug camera. The rotational measuring procedure generates Scheimpflug images in three dimensions.
- group high myopia (Experimental): 1. Patients with high myopia aging more than 15 years old
  2. All patients are with visual acuity (uncorrected, with habitual correction, and best spectacle correction).
  3. There is no restrictions on the range and regularity of keratometry
  Interventions: Diagnostic Test: Using Oculus Pentacam® which is s a rotating Scheimpflug camera. The rotational measuring procedure generates Scheimpflug images in three dimensions.
- group Hypermetropia (Experimental): 1. Patients with hypermetropia aging more than 15 years old
  2. All patients are with visual acuity (uncorrected, with habitual correction, and best spectacle correction).
  3. There is no restrictions on the range and regularity of keratometry
  Interventions: Diagnostic Test: Using Oculus Pentacam® which is s a rotating Scheimpflug camera. The rotational measuring procedure generates Scheimpflug images in three dimensions.
- group mixed astigmatism (Experimental): 1. Patients with mixed astigmatism aging more than 15 years old
  2. All patients are with visual acuity (uncorrected, with habitual correction, and best spectacle correction).
  3. There is no restrictions on the range and regularity of keratometry
  Interventions: Diagnostic Test: Using Oculus Pentacam® which is s a rotating Scheimpflug camera. The rotational measuring procedure generates Scheimpflug images in three dimensions.

INTERVENTIONS:
Diagnostic Test: Using Oculus Pentacam® which is s a rotating Scheimpflug camera. The rotational measuring procedure generates Scheimpflug images in three dimensions. — Scheimpflug imaging attains a wide and high depth-of-focus , providing sharp images that include information from an anterior corneal surface through to the posterior crystalline capsule
  Other Names: The scheimpflug principle describes the optical imaging condition

SUMMARY:
To evaluate corneal topographic pattern & its correlation with refractive status of the eye .

DETAILED DESCRIPTION:
This study will be established in The Future Center for refractive surgery, Sohag, Egypt.

This study will include 100 eyes of patients aged over 15 years. All patients were subjected to topography imaging.

Using Oculus Pentacam® which is s a rotating Scheimpflug camera. The rotational measuring procedure generates Scheimpflug images in three dimensions.

The scheimpflug principle describes the optical imaging condition when the plane of an object is not parallel to the film of the camera and has to cut each other in one line or one point of intersection with the advantage to achieve wide depth of focus.

Scheimpflug imaging attains a wide and high depth-of-focus , providing sharp images that include information from an anterior corneal surface through to the posterior crystalline capsule; this depends mainly on media transparency and pupil size .

ELIGIBILITY:
Inclusion Criteria:

* Patients aging more than 15 years old
* All patients are with visual acuity (uncorrected, with habitual correction, and best spectacle correction).
* There is no restrictions on the range and regularity of keratometry.

Exclusion Criteria:

* Patients with a history of any trauma to the eye.
* Patients with recent contact lens wear.
* history of ocular surgery .
* Patients with distance corrected visual acuity or abnormal retinoscopy examination (e.g., scissoring reflex).

  5. If there was any error in reading the topographic map. 6. Patients with anemotropic refraction.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Thickness | 3 months after begin of study
  Topographic values using Oculus Pentacam®
degree of astigmatism in D | 3 months after begin of study
  Topographic values using Oculus Pentacam®
maximum keratometry | 3 months after begin of study
  Topographic values using Oculus Pentacam®
front and back elevation of the apex (um). | 3 months after begin of study
  Topographic values using Oculus Pentacam®

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Iqbal, MD.PhD, Study Chair — Sohag Faculty of medicine
Locations (1):
- Facultyof medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT05626075/Prot_000.pdf